CLINICAL TRIAL: NCT07289451
Title: TLR 9 (rs352140) Gene Polymorphism in Helicobacter Pylori Infection in Children
Brief Title: TLR 9 (rs352140) Gene Polymorphism in Helicobacter Pylori Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Nashwa farouk Mohamed, lecturer of pediatrics, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MS-14-12-2022
Record Dates: First submitted 2025-11-25; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: H. Pylori Infection
Keywords: TLR 9
MeSH Terms: interventions — Polymorphism, Genetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- children with age between 1 and 18 years with gastrointestinal symptoms that necessitates upper dige (Experimental): children with age between 1 and 18 years with gastrointestinal symptoms that necessitates upper digestive endoscopy like: persistent pain in the abdomen and/or the stomach, Heartburn, vomiting, and nausea.
  Additionally, children who showed red flag signs like anemia, gastrointestinal hemorrhage, failure to thrive, or increased ESR were as well involved.
  Interventions: Diagnostic Test: TLR TLR 9 (rs352140) gene polymorphism

INTERVENTIONS:
Diagnostic Test: TLR TLR 9 (rs352140) gene polymorphism — Genotyping of TLR9 (rs352140) was done using TaqMan mechanism on the Applied Biosystems™ 7500Fast Dx Real-Time PCR System (Applied Biosystems, Waltham, MA, United States) and a predesigned assay, namely C_2301954_20.
  A venous blood sample (2 mls) were withdrawn from each subject and were collected into sterile ethylene diaminetetra acetate "EDTA" (vacutainer) tube and were used for DNA extraction. DNA was extracted from fresh samples and stored at -20 °C till time of assay for determination of TLR9 (rs352140) polymorphism by using real time Polymerase chain reaction (rt PCR) technique. The blood samples were used for DNA extraction using the Gene JET Whole Blood Genomic DNA purification Mini Kit (Thermo Fisher Scientific, Germany) according to the manufacturer's protocol. Determination of DNA concentration was done using Nanodrop One spectrophotometer (thermoscientific, USA). A concentration of (1µg) from each sample was used for genotyping by rtPCR assay. Genotyping of TLR9 (rs352140)

SUMMARY:
study aimed to identify the role of TLR9 (rs352140) gene in suppressing or promoting the inflammation related to H. pylori infection in children.This cross-sectional study was conducted on 50 children with positive H. pylori infection and 50 age and sex matched, negative H. pylori children, all children undertook full history, complete clinical investigation, laboratory testing, upper digestive endoscopies and genotyping of TLR9 (rs352140).

DETAILED DESCRIPTION:
H. pylori infection is acknowledged as one of the major causes of gastrointestinal bacterial infections globally, imposing a substantial load on public health organizations, mostly in low-resource countries . H. pylori infection continues to pose a substantial challenge, particularly in vulnerable populations like infants, despite the significant advance made in health care organization and medicine .

The implications of H. pylori infection in minors have a profound impact on numerous aspects of health and well-being, which extend beyond the gastrointestinal tract.

In addition to its immediate effect on the gastric mucosa integrity of, H. pylori infection has systemic impacts that can have a negative impact on, growth trajectories, the nutritional status and overall health results of children who are affected .

A variety of gastrointestinal disorders, involving moderate gastritis and additional serious diseases like peptic ulcer disease, have been correlated with chronic infection by H. pylori. In addition, epidemiologic evidence indicates a potential correlation between an elevated hazard for acquiring gastric adenocarcinoma and mucosa-associated lymphoid tissue lymphoma in later life and the acquisition of H. pylori infection during childhood. These long-term effects reinforce the urgent need to address H. pylori infection in children as a major community health importance .

Currently, there are numerous invasive and non-invasive diagnostic assessments accessible to identify H. pylori infection in children. However, tissue culture and the rapid urease test or concordant-positive histopathology tests remains the gold standard results .

Mast, macrophages, dendritic, eosinophils, neutrophils, and natural killer (NK) cells are cell actors of the innate immune system which provide antigen-independent defense against H. pylori infection .

Toll-like receptors (TLRs) are critical innate immunity regulators that can be stimulated upon the identifying of pathogen-associated molecular patterns (PAMPs) such as viral and bacterial ligands. They serve as the initial line of defense for the host against a variety of circumstances, involving H. pylori infection .

There are 13 TLRs (TLR1-13) in mammals, but only 10 (TLR1-10) are present in humans, but all are present in mice, with TLR10 being nonfunctional.

The human stomach's gastric epithelial cells are known to produce TLR4 and TLR9, which are crucial for innate immune signaling to H. pylori .

ELIGIBILITY:
Inclusion Criteria:

1. children with age between 1 and 18 years with gastrointestinal symptoms that necessitates upper digestive endoscopy like:

   * persistent pain in the abdomen and/or the stomach,
   * Heartburn,
   * vomiting,
   * nausea.
2. children who showed red flag signs like :

   * anemia,
   * gastrointestinal hemorrhage,
   * failure to thrive,
   * increased ESR .

Exclusion Criteria:

* cases on proton pump inhibitors,
* those with substantial medical diseases,
* those with gastrointestinal conditions that could explain their stomach discomfort (such as celiac disease, functional abdominal pain and inflammatory bowel disease).

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
TLR9 rs352140 gene polymorphism correlation with of H. pylori infection and incidence of gastritis in children | in 1 to 3 months of complaint
  determination of TLR9 (rs352140) polymorphism by using real time Polymerase chain reaction (rt PCR) technique
TLR9 rs352140 gene polymorphism with abdominal pain , H. pylori infection and incidence of gastritis in children | in 1 -3months of symptoms
  determination of TLR9 (rs352140) polymorphism by using real time Polymerase chain reaction (rt PCR) technique

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Benha University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wicherska-Pawlowska K, Wrobel T, Rybka J. Toll-Like Receptors (TLRs), NOD-Like Receptors (NLRs), and RIG-I-Like Receptors (RLRs) in Innate Immunity. TLRs, NLRs, and RLRs Ligands as Immunotherapeutic Agents for Hematopoietic Diseases. Int J Mol Sci. 2021 Dec 13;22(24):13397. doi: 10.3390/ijms222413397. PMID 34948194
- [Result] Elbehiry A, Marzouk E, Aldubaib M, Abalkhail A, Anagreyyah S, Anajirih N, Almuzaini AM, Rawway M, Alfadhel A, Draz A, Abu-Okail A. Helicobacter pylori Infection: Current Status and Future Prospects on Diagnostic, Therapeutic and Control Challenges. Antibiotics (Basel). 2023 Jan 17;12(2):191. doi: 10.3390/antibiotics12020191. PMID 36830102
- [Result] Nguyen J, Kotilea K, Bontems P, Miendje Deyi VY. Helicobacter pylori Infections in Children. Antibiotics (Basel). 2023 Sep 12;12(9):1440. doi: 10.3390/antibiotics12091440. PMID 37760736